CLINICAL TRIAL: NCT04211285
Title: e-GAB: Electronic Geriatric Assessment Bundle: Development of an Arabic Self-administered Android CGA Application
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Doha Rasheedy, Assistant Professor of Geriatric Medicine, Ain Shams University
Other Study IDs: AinShamsUGer
Record Dates: First submitted 2019-01-23; First posted 2019-12-26 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Health Services for the Aged; Frailty; Cognitive Impairment; Depression; Disability Physical; Urinary Incontinence; Malnutrition
Keywords: comprehensive geriatric assessment; telemedicine; multidisciplinary approach of elderly care; electronic geriatric assessment bundle
MeSH Terms: conditions — Frailty; Cognitive Dysfunction; Depression; Urinary Incontinence; Malnutrition

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- community dwelling elderly: community dwelling elderly patients (60 years or older), can read and write, able to use the android software applications
  Interventions: Diagnostic Test: e-GAB; Diagnostic Test: standard physician performed CGA

INTERVENTIONS:
Diagnostic Test: e-GAB — android application for comprehensive geriatric assessment
Diagnostic Test: standard physician performed CGA — CGA by an experienced geriatrician blinded to the result of e-GAB

SUMMARY:
The aim of this study is to design and assess the accuracy of administering the electronic Geriatric Assessment Bundle (e-GAB) compared to geriatrician performed comprehensive geriatric assessment (CGA) in a group of Egyptian elderly. The development of an Arabic software platform for CGA can improve the clinical practice by providing a valid user friendly tool to collect and analyze data for geriatric patients attending non- Geriatric health care service.

DETAILED DESCRIPTION:
Modern geriatric care is based primarily on the concept of multidisciplinary approach of elderly care. This could be achieved by integrating CGA in different disciplines dealing with the older patient. CGA is different from that of the standard medical evaluation; it is a systematic evaluation of frail older adults. It uses combinations of validated geriatric tools to formulate an inventory of health problems, and develop an individualized geriatric intervention plan.

The software platform for CGA has been widely used in western countries; however, tools that can fit patients with different backgrounds should be implemented..

From the initial pool of 3 potential subtests, four experienced geriatricians developed a bundle of 15 subtests, to evaluate cognition, mood, vision, hearing, urinary continence, nutrition, functional capacity, fall risk and balance impairment, frailty, polypharmacy, sleep, pain, home safety, and social problems. Moreover, a rapid survey of medical and surgical conditions was obtained.

Initial evaluation of these subsets compared to the reference standard CGA was done. Each patient completed the bundle then underwent CGA by an experienced geriatrician blinded to the result of e-GAB

ELIGIBILITY:
Inclusion Criteria:

* 60 years or above
* community dwelling
* can read and write
* can use the android application

Exclusion Criteria:

* any patient refused to participate

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 50 elderly patients completed the bundle then underwent CGA by an experienced geriatrician blinded to the result of e-GAB
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
the sensitivity and specificity of administering the electronic Geriatric Assessment Bundle (e-GAB) | the geriatrician will perform standard CGA within 30 minutes of e-GAB completion
  assess sensitivity and specificity of the e-GAB for detecting the aforementioned conditions (e.g. Frailty, Depression, sleep disturbance, malnutrition, cognitive decline etc.. )compared to standard CGA

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt